CLINICAL TRIAL: NCT06496672
Title: The Wrist-Free Study- A Randomized Controlled Trial Comparing Traditional Above Elbow Casts to Ones That Free the Wrist in Pediatric Supracondylar Humerus Fractures
Brief Title: The Wrist-Free Study - Comparing Traditional Above Elbow Casts to Ones That Free the Wrist
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KKWCHWristFree
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Supracondylar Humerus Fracture
Keywords: Pediatric

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional (Active Comparator): Participants in this group receive the existing treatment, which is a cast that terminates at the palmar bar.
  Interventions: Procedure: Traditional long arm cast
- Modified (Experimental): Participants in this group receive the experimental treatment, a cast that terminates at the wrist.
  Interventions: Procedure: Modified long arm cast

INTERVENTIONS:
Procedure: Modified long arm cast — A shorter cast that frees the wrist
  Arms: Modified
Procedure: Traditional long arm cast — Current standard of care where the cast extends up to the palmar bar
  Arms: Traditional

SUMMARY:
This randomized controlled trial compares clinical outcomes, patient comfort and satisfaction of freeing the wrist in casts for supracondylar humerus fractures in children.

ELIGIBILITY:
Inclusion Criteria:

* Type I and Type IIa Supracondylar Humerus Fracture

Exclusion Criteria:

* History of elbow injury
* Polytrauma

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | 3-4 Weeks
  Measured using QDASH

SECONDARY OUTCOMES:
Complications in healing | 3-4 Weeks
  Observe for loss of reduction in fracture

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth PL Wong, FRCS, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khoshbin A, Leroux T, Wasserstein D, Wolfstadt J, Law PW, Mahomed N, Wright JG. The epidemiology of paediatric supracondylar fracture fixation: a population-based study. Injury. 2014 Apr;45(4):701-8. doi: 10.1016/j.injury.2013.10.004. Epub 2013 Oct 17. PMID 24183392
- [Background] Micheloni GM, Novi M, Leigheb M, Giorgini A, Porcellini G, Tarallo L. Supracondylar fractures in children: management and treatment. Acta Biomed. 2021 Jul 26;92(S3):e2021015. doi: 10.23750/abm.v92iS3.11725. PMID 34313666
- [Background] Boyd AS, Benjamin HJ, Asplund C. Splints and casts: indications and methods. Am Fam Physician. 2009 Sep 1;80(5):491-9. PMID 19725490
- [Background] Shenoy PM, Islam A, Puri R. Current Management of Paediatric Supracondylar Fractures of the Humerus. Cureus. 2020 May 15;12(5):e8137. doi: 10.7759/cureus.8137. PMID 32550057
- [Background] Vaquero-Picado A, Gonzalez-Moran G, Moraleda L. Management of supracondylar fractures of the humerus in children. EFORT Open Rev. 2018 Oct 1;3(10):526-540. doi: 10.1302/2058-5241.3.170049. eCollection 2018 Oct. PMID 30662761